CLINICAL TRIAL: NCT03065114
Title: Institute of Medicine, Chung Shan Medical University
Brief Title: Retrospective Study on Clinical Results of Preimplantation Genetic Screening at Different Embryo Stage
Status: Completed | Type: Observational
Sponsor: Yeh (Other)
Responsible Party: Sponsor-Investigator, Yeh, Institutional Review Board of Chung Shan Medical University, Chung Shan Medical University
Organization: Chung Shan Medical University (Other)
Other Study IDs: CS14124
Record Dates: First submitted 2017-02-22; First posted 2017-02-27 (Actual); Last update posted 2017-02-27 (Actual); Status verified 2017-02

CONDITIONS: Genetic Disorder; Fertility Disorders; Reproductive Disorder
MeSH Terms: conditions — Genetic Diseases, Inborn

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PGSno.: blastocysts from patients underwent preimplantational genetic screen (PGS) prtocols. only euploid embryos were selected to transfer.
  Interventions: Other: PGS

INTERVENTIONS:
Other: PGS — chromosome abnormality test from PGS and relationship between embryo development

SUMMARY:
Preimplantational genetic screen (PGS) is tool for diagnosis of embryo chromosome abnormality before transfer. Under this tool, patients with a family history of genetic disease or special genetic disease could avoid to produce chromosomal abnormalities of the next pregnant. This study is a retrospective study, data collection from 2001 Jan. to 2015. Nov. Patients underwent PGS and data including the couples age, infertility factors, stimulation protocols, medicine records, embryo quality records and blood tests were collected in this study. Analysis the relationship between outcomes of PGS, clinical outcomes and embryo quality is performed and further to find a diagnosis reference for clinical care.

DETAILED DESCRIPTION:
Research background Preimplantational genetic screen (PGS) is tool for diagnosis of embryo chromosome abnormality before transfer. Under this tool, patients with a family history of genetic disease or special genetic disease could avoid to produce chromosomal abnormalities of the next pregnant. For the preemergence of embryos before the genetic diagnosis must be carried out artificial reproductive treatment, the process includes induction of ovulation, ovulation, in vitro fertilization and embryo culture, to embryos grow to six to eight cells or cultured into the stage of blastocyst stage, Under the embryonic section, take one or several cells, the slices of cells for genetic diagnosis, select the embryo without genetic disease implanted in the uterine cavity, in order to avoid the birth of genetic disease offspring.

PGS can reduce the pregnancy when the chromosomal abnormalities of the fetus after implantation, but also to reduce the risk of abortion from chromosomal abnormalities, and can avoid the couples implanted with genetic abnormalities of the embryos, thereby significantly reducing it is important to promote the process of eugenics and reduce the social cost.

Research purposes The detection of chromosomal abnormalities of embryos are important factors for clinical diagnosis or screening before implantation. However, there is no complete analysis of domestic studies. This program will compare the genes or chromosomal abnormalities and clinical outcomes of embryo testing at different stages of embryonic development.

Research design This study is a retrospective study, data collection from 2001 Jan. to 2015. Nov. Patients underwent PGS and data including the couples age, infertility factors, stimulation protocols, medicine records, embryo quality records and blood tests were collected in this study. Analysis the relationship between outcomes of PGS, clinical outcomes and embryo quality is performed and further to find a diagnosis reference for clinical care.

ELIGIBILITY:
Inclusion Criteria:

* Women underwent in vitro fertilization (IVF) treatment and preimplantational genetic screen (PGS).

Exclusion Criteria:

* N/A

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women underwent in vitro fertilization (IVF) treatment and preimplantational genetic screen (PGS).
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2014-12-01 (Actual); Primary Completion 2015-11-30 (Actual); Study Completion 2015-11-30 (Actual)

PRIMARY OUTCOMES:
implantation rate | 1~2 week after pregnancy test
  detection sac after embryo transfer

CONTACTS AND LOCATIONS:
Overall Officials: Maw-Sheng Lee, Phd, Study Chair — Lee's Women Hospital

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Chen HH, Huang CC, Cheng EH, Lee TH, Chien LF, Lee MS. Optimal timing of blastocyst vitrification after trophectoderm biopsy for preimplantation genetic screening. PLoS One. 2017 Oct 5;12(10):e0185747. doi: 10.1371/journal.pone.0185747. eCollection 2017. PMID 28982142